CLINICAL TRIAL: NCT04203875
Title: Abatacept for Treatment of Recurrent or de Novo Autoimmune Hepatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of eligible study participants.
Sponsor: Stuart Knechtle, M.D. (Other)
Responsible Party: Sponsor-Investigator, Stuart Knechtle, M.D., Transplant Surgeon, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102357
Record Dates: First submitted 2019-12-12; First posted 2019-12-18 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Abatacept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Orencia® (Abatacept) (Experimental): Abatacept 125 mg, subcutaneous once a week for 6 months or up to one year if subject has a favorable response
  Interventions: Drug: Orencia® (Abatacept)

INTERVENTIONS:
Drug: Orencia® (Abatacept) — Orencia® (Abatacept) will be administered once a week for 6 months subcutaneously (injection under the skin) with an option to continue to receive Abatacept weekly injections for an additional 6 months, for a total of 12 months if there is a positive response.

SUMMARY:
The purpose of this study is to evaluate whether Orencia® (Abatacept) improves outcomes in liver transplant patients with recurrent or de novo AIH (autoimmune hepatitis) that has not responded to previous therapy. AIH that does not respond to steroids or conventional immunotherapy often affects young patients and leads to irreversible liver damage. There is currently no effective therapy for this condition.

DETAILED DESCRIPTION:
Participants in this study will receive the study drug once a week for 6 months. If the study doctor feels the study drug has been beneficial, participants may receive additional study drug doses for up to an additional 6 months. Participants will continue on follow-up for 1 year after stopping Abatacept.

The risks related to participation in this study include potential side effects from the study drug include infusion-related reactions (reactions at the injection site), increase in respiratory adverse events, infections in patients with chronic obstructive pulmonary disease, risk of development of malignancies (cancer) or autoimmune disorders (which may make your current autoimmune disease worse or you can contract new autoimmune diseases). It is unknown if this is drug related. The study doctor will discuss any concerns about this with you prior to receiving treatment.

There is the possibility that the participant may experience improvement in their medical condition from participation in this study. However, this benefit cannot be guaranteed. There may be no direct medical benefit to the participant due to their participation. The Investigator hopes that in the future the information learned from this study will benefit other people with this condition.

ELIGIBILITY:
Inclusion Criteria for de novo AIH

* Age 18 or older
* Patients who have biopsy evidence of autoimmune liver disease following liver transplantation and a different pre-transplant etiology of liver disease will be eligible.
* Patients who have been treated with steroids or other immunosuppressive agents for at least a month and who have not responded either with respect to normalization of liver function tests or biopsy evidence of hepatitis will be eligible.
* Ability to provide signed and dated IRB approved written consent in accordance with regulatory and institutional guidelines prior to any protocol-related procedure.
* Women of child bearing potential agree to have pregnancy test at screening
* Males agree use of appropriate contraceptives during the active Orenia dosing period

Inclusion Criteria for recurrent AIH

* Age 18 or older
* Patients who have biopsy evidence of autoimmune liver disease following liver transplantation and whose original etiology of liver disease was AIH will be eligible.
* Patients who have been treated with steroids or other immunosuppressive agents for at least a month and who have not responded either with respect to normalization of liver function tests or biopsy evidence of hepatitis will be eligible.
* Ability to provide signed and dated IRB approved written consent in accordance with regulatory and institutional guidelines prior to any protocol-related procedure.
* Women of child bearing potential agree to have pregnancy test at screening
* Males agree use of appropriate contraceptives during the active Orenia dosing period

Exclusion Criteria:

* Active systemic infection
* Allergy to abatacept
* Known malignancy in the previous 2 years except for non-melanoma skin cancer
* Pregnancy or breast feeding
* Inability to commit to complete treatment protocol at Duke, as all procedures must be completed at Duke
* Prisoners or those who are compulsory detained
* Inability to read and understand English
* EBV seronegative (if not tested within 2 years prior to study enrollment, then testing will be done prior to study enrollment, results must be positive for study participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events as reported | within 56 days of last dose
  Any Adverse Event
Number of Infections seen after administration | within 56 days of last dose
  Any infection
Number of malignancies reported | within 56 days of last dose
  any malignancy

SECONDARY OUTCOMES:
A change in aspartate aminotransferase (AST) | Baseline and at 6 weeks after start of administration
  Any change
A change in alanine aminotransferase (ALT) | Baseline and at 6 weeks after start of administration
  Any change
a change in alkaline phosphatase | Baseline and at 6 weeks after start of administration
  Any change
Change in bilirubin | Baseline and at 6 weeks after start of administration
  Any change
Change in liver biopsy evidence of AIH compared to pre-treatment | through study completion, an average of 1 year
  evidence of worsening AIH on biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Knechtle, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD at this time